CLINICAL TRIAL: NCT03799692
Title: Clinical Trial of Nanoparticle Albumin-Bound Paclitaxel Combined With Carboplatin as Neoadjuvant Chemotherapy in Luminal B/HER-2 Negative Breast Cancer
Brief Title: Albumin-Bound Paclitaxel Combined With Carboplatin as Neoadjuvant Chemotherapy in Luminal B/HER-2 Negative Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1808189-8
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: HER-2 Negative Breast Cancer
Keywords: Neoadjuvant Chemotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Experimental): Nanoparticle Albumin-Bound Paclitaxel 125mg/m2, iv, Carboplatin AUC=2, iv, d1, 8, 15, 4 cycles (21 days per cycle).
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Drug: Nanoparticle Albumin-Bound Paclitaxel Nanoparticle Albumin-Bound Paclitaxel 125mg/m2, iv, d1, 8, 15.
  Drug: Carboplatin AUC=2 iv, d1, 8, 15.

SUMMARY:
This is an open-label, single arm, two-stage Simon Design study for women with LuminalB/HER-2 Negative Breast Cancer treated with Nanoparticle Albumin-Bound Paclitaxel and Carboplatin.

The primary objective of the trial is to evaluate of the efficacy and safety of Nanoparticle Albumin-Bound Paclitaxel Combined with Carboplatin as Neoadjuvant Chemotherapy in Luminal B/HER-2 Negative Breast Cancer.

The primary endpoint of the study is to assess Pathological complete response rate（pCR）using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

The total number of patients to be included in this study is 78 patients.

The duration of the study, from first patient visit to last patient visit will be approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age: from 18 to 70 years old, female.
* 2.Has histologically or cytologically confirmed unilateral primary invasive breast cancer with a clinical stage of T2-4NanyM0.
* 3.Immunohistochemical detection of ER+, PR+, HER-2 negative (if HER2 expression is 2+ patients need to be confirmed by in situ hybridization to detect no HER-2 gene amplification) and Ki-67 expression >20% of patients;
* 4.At least one measurable objective lesion according to RECIST 1.1 criteria.
* 5.ECOG performance status of 0-1.
* 6.Bone marrow function: Neutrophils ≥ 1.5×109/L, platelets ≥ 100×109/L, and hemoglobin ≥ 90 g/L.
* 7.Liver and renal function: Serum creatinine ≤ 1.5 times the upper limit of normal. AST and ALT ≤ 2.5 times the upper limit of normal Total bilirubin ≤ 1.5 times the upper limit of normal, or ≤ 2.5 times the upper limit of normal in patients with Gilbert's syndrome.
* 8.Has good compliance with the planned treatment, understand the study process and sign written informed consent.

Exclusion Criteria:

* 1.Any prior cytotoxic chemotherapy, endocrine therapy, biological therapy, or radiation therapy.
* 2.Patients with grade II or higher heart disease scored by the New York Heart Association (NYHA).
* 3.Severe systemic infection, or with other serious diseases.
* 4.Patients with known hypersensitivity or intolerance to chemotherapeutic agents or their excipients.
* 5.Other malignancies have occurred in the past 5 years, except for cured cervical carcinoma in situ, non-melanoma skin carcinoma.
* 6.Pregnant or lactating, and who refuse to take appropriate contraception during the course of this trial.
* 7.Have participated in other study studies within 30 days prior to the first dose of study drug.
* 8.Patients who, in the opinion of the Investigator, are not suitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is pathological complete remission (pCR) | 3 months
  Histopathological examination of breast and axillary lymph node specimens without invasive cancer cell remnants. Complete pathological response is also considered to be achieved if only in situ cancer cell remnants are present in the surgical specimens.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 3 months
  The second endpoint ORR composed of tumor response classifications of complete response (CR) and partial response (PR), refers to the number of cases with complete and partial response after treatment as a percentage of the total number of evaluable cases.
Breast conserving surgery (BCS) rate | 3 months
  Percentage of patients undergoing breast-conserving surgery after neoadjuvant therapy as a whole evaluable.
Adverse events (AE) | 3 months
  Adverse events (AE) were monitored on an ongoing basis and classified according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03. Patients were assessed for toxicities before each administration, and toxicity was graded accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Department of Breast Surgery, Cancer Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided